CLINICAL TRIAL: NCT00356291
Title: HIV Prevention for the Mentally Ill: Motivation-Skills
Brief Title: Improving HIV Prevention Skills in People With Serious Mental Illnesses
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Stephen Brady, Director, Mental Health Counseling & Behavioral Medicine Program Associate Professor of Psychiatry Boston University School of Medicine, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34MH075644 (NIH); R34MH075644 (NIH); DAHBR 9A-ASNM
Record Dates: First submitted 2006-07-21; First posted 2006-07-25 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: HIV/AIDS
Keywords: HIV; AIDS; Prevention; Serious Mental Illness
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

ARMS (2):
- 1 (Experimental): Participants will receive Skill-Building and Motivational Interviewing.
  Interventions: Behavioral: Skill-Building (SB) plus Motivational Interviewing
- 2 (Active Comparator): Participants will receive Skill-Building.
  Interventions: Behavioral: Skill-Building (SB)

INTERVENTIONS:
Behavioral: Skill-Building (SB) plus Motivational Interviewing — SB is a 4 to 5 session individually-based psychoeducational intervention. Participants meet weekly with an interventionist for 3 to 4 weeks and then receive a booster session 3 months after baseline. The traditional Skill-Building intervention will be augmented with Motivational Interviewing techniques.
  Arms: 1
Behavioral: Skill-Building (SB) — SB is a 4-session individually-based psychoeducational HIV risk reduction intervention. Participants meet weekly with an interventionist for 3 weeks and then receive a booster session 3 months after baseline.
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of motivational interviewing plus skill building in reducing HIV risk behavior in people with serious mental illnesses.

DETAILED DESCRIPTION:
People with serious mental illness (SMI) are at higher risk for contracting HIV than the general population. Although fewer people with SMI are sexually active, as compared to the healthy population, those with SMI who are sexually active tend to engage in sexual behaviors that put them at increased risk for HIV and other STDs. The onset of SMI, which often interferes with normal psychosocial development, may cause these behaviors. Additionally, SMI is frequently associated with poor judgment, affective instability, and impulsiveness. Interventions designed to reduce the risk for contracting HIV in people with SMI exist, but they have had little success. New approaches to treating this population are essential. This study will evaluate the effectiveness of motivational interviewing (MI) plus skill building (SB) exercises in reducing HIV risk behavior in people with SMI.

Participants in this 6-month, open-label study are randomly assigned to partake in SB training either alone or combined with MI. The skill building program focuses on behavioral skills training, with an emphasis on negotiating and communicating with prospective partners. Training includes information about HIV risk, including mechanisms of transmission, abstinence, and safer sex and drug use behaviors; HIV risk reduction strategies, including condom use, abstinence/safer sex negotiation skills, and reduced/safer drug use; and an opportunity to be tested for HIV if the participant has not already done so. The SB plus MI intervention (SB-MI) includes components of the SB intervention, as well as elements of MI. MI includes identifying high risk sexual and drug use behaviors related to HIV; reducing the ambivalence about making high risk behavior changes; increasing motivation to change high risk behaviors; and developing a plan to implement these changes. HIV testing may be included. Participants in both interventions report to the study site on six to seven occasions over the course of the study. The visits last between 1 and 2 hours and include both treatment and evaluation. Participants attend two follow-up visits, one 3 months after randomization, and one 6 months after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for a serious and persistent mental illness (as defined by the Massachusetts Department of Mental Health)
* English-speaking
* Engagement in HIV risk behavior within 3 months prior to study entry
* Ability to keep study-related appointments

Exclusion Criteria:

* Unstable mental status

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2007-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Timeline Followback (TLFB) measures of HIV risk behaviors and use of HIV risk prevention strategies (including use of male and female condoms, dental dams, and recommended intravenous needle-cleaning) | Measured at Months 3 and 6
Communication and negotiation skills | Measured at Months 3 and 6
Simulated demonstrations of use of male and female condoms, dental dams, and intravenous needle cleaning | Measured at Months 3 and 6
Access of HIV counseling and testing | Measured at Months 3 and 6

SECONDARY OUTCOMES:
HIV knowledge (HIV/AIDS Knowledge Questionnaire - HIV-KQ) | Measured at Months 3 and 6
Multidimensional Condom Attitude Scale (MCAS) | Measured at Months 3 and 6

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M. Brady, PhD, Principal Investigator — Boston University
Locations (1):
- Boston University Medical Center, Boston, Massachusetts, United States